CLINICAL TRIAL: NCT02943226
Title: IV Contrast Administration: Effect of Three Side Hole Infusion Catheter on CT Image Quality, Infusion Pressure, and Infusion Rates, Compared to a Standard Infusion Catheter
Brief Title: Effect of Three Side Hole Infusion Catheter on CT Image Quality Compared to a Standard Infusion Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Joseph P Hasapes, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: HSC-MS15-0906
Record Dates: First submitted 2016-10-20; First posted 2016-10-24 (Estimated); Results first posted 2018-02-12 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Contrast Enhanced Computed Tomography (CT) Scanning

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Becton Dickinson Nexiva Diffusics System (Experimental): Intervention with the new Becton Dickinson Nexiva Diffusics System will be evaluated to see if it will improve image quality compared to the standard catheter.
  Interventions: Device: Becton Dickinson Nexiva Diffusics System
- Standard intravenous catheter (Active Comparator): Standard catheter with one hole at the tip will be compared to novel 3 hole Becton Dickinson Nexiva Diffusics System to see which catheter provides the best image quality.
  Interventions: Device: Standard intravenous catheter

INTERVENTIONS:
Device: Becton Dickinson Nexiva Diffusics System — Becton Dickinson Nexiva Diffusics System will be used to inject IV contrast and will be compared to a single hole catheter to see if it improves image quality in the main vessels in the abdomen and pelvis because of its novel design.
  Arms: Becton Dickinson Nexiva Diffusics System
Device: Standard intravenous catheter — Standard catheter with one hole at the tip will be compared to a novel 3 hole catheter to see which catheter provides the best image quality.
  Arms: Standard intravenous catheter

SUMMARY:
The purpose of this research study is to compare two types of catheters used for infusing the contrast dye necessary for viewing internal organs during computed tomography (CT) scanning. The standard catheter, which has one hole from which contrast dye enters veins, will be compared to the Becton Dickinson Nexiva Diffusics System catheter, which has three holes for diffusing dye into veins. The purpose of this study is to determine which catheter type gives the best image.

DETAILED DESCRIPTION:
This will be a prospective, randomized, controlled trial. The catheter is already in use at our facilities. After informed consent, patients will be randomly given the standard or new catheter in our practice. Envelopes with the random assignment will be available to the individuals consenting patients. Randomization generally ensures that study groups are similar on average. As age, sex, and weight impact image quality, we will collect data on these factors in case randomization results in an imbalance. This will allow for control of these factors in analysis of the data. Data will be collected from CT abdomen pelvis examinations within a 6 month-1 year period in 2016 - 2017. Our primary outcome is image quality, measured as tissue density and distribution of contrast within the liver, spleen, aorta and IVC. Our secondary outcomes include Peak Contrast Infusion Pressure and Injection Flow Rate. Possible adverse events for use of any type of catheter include contrast infiltration into the subcutaneous tissues which is a minor limited event. All infiltrations will be recorded as part of the permanent medical record, documented in the chart, and the referring physician notified. The patient will be assessed by a physician immediately and referred to the ED if necessary for further evaluation. Current technology utilizes Power injector equipment which alerts the technologist to the pressure being achieved. If the injection pressure exceeds 325 psi the Power injector automatically shuts off.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing contrast enhanced CT abdomen pelvis examinations at Lyndon B. Johnson General Hospital in Texas
* Patients whose access point is the antecubital fossa
* Patients receiving 20 or 22 gauge catheters for their CT exam
* Patients scanned on two 64 slice CT scanners at the same hospital

Exclusion Criteria:

* patients whose access point is other than antecubital fossa

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Hasapes, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Becton Dickinson Nexiva Diffusics System Fenestrated Catheter: Becton Dickinson (BD) Nexiva™ Diffusics™ System uses three laser-cut tear-drop holes located in the catheter tip to stabilize the catheter tip by reducing flow velocities while maintaining flow rates during intravenous contrast administration into the vein.
- Standard Intravenous Non-fenestrated Catheter: The standard catheter has one hole at the tip for contrast infusion.
Period: Overall Study
Arm/Group | Becton Dickinson Nexiva Diffusics System Fenestrated Catheter | Standard Intravenous Non-fenestrated Catheter
Started | 31 | 30
Completed | 31 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Becton Dickinson Nexiva Diffusics System Fenestrated Catheter | Standard Intravenous Non-fenestrated Catheter | Total
Number analyzed (Participants) | 31 | 30 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (11.2) | 52.9 (13.8) | 51.9 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 33
  Male | 15 | 13 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 31 | 30 | 61
Abdominal anterioposterior diameter at lower kidneys [Mean (Standard Deviation); unit: centimeters] | 27.0 (5.1) | 26.6 (4.4) | 26.8 (4.7)
Abdominal transverse (left-right) diameter at lower kidneys [Mean (Standard Deviation); unit: centimeters] — Population: Abdominal transverse (left-right) diameter at lower kidney data was not collected for all subjects.
  centimeters
    number analyzed (Participants) | 29 | 29 | 58
    (all) | 38.7 (7.9) | 37.0 (5.7) | 37.1 (6.1)

OUTCOME MEASURES:

1. Primary Outcome: Image Quality as Assessed by Ratio of Tissue Density of Main Portal Vein (MPV) to the Aorta
Description: The ratio of tissue density measured in the main portal vein (MPV) to tissue density in the aorta on the CT images will be determined and will provide a measure of biodistribution, which is an important indicator of image quality. Dividing each Hounsfield unit measurement by the aorta density and determining these ratios will be done on a per patient basis to assess biodistribution as a measure of image quality.
Time Frame: at the time of CT scanning
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Becton Dickinson Nexiva Diffusics System Fenestrated Catheter | Standard Intravenous Non-fenestrated Catheter
Number analyzed (Participants) | 31 | 30
Ratio | 0.95 (0.18) | 0.95 (0.18)

2. Primary Outcome: Image Quality as Assessed by Ratio of Tissue Density of Spleen to the Aorta
Description: The ratio of tissue density measured in the spleen to tissue density in the aorta on the CT images will be determined and will provide a measure of biodistribution, which is an important indicator of image quality. Dividing each Hounsfield unit measurement by the aorta density and determining these ratios will be done on a per patient basis to assess biodistribution as a measure of image quality.
Time Frame: at the time of CT scanning
Population: Data for the "Becton Dickinson Nexiva Diffusics System fenestrated catheter" arm was not collected for one patient because the patient had a splenectomy.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Becton Dickinson Nexiva Diffusics System Fenestrated Catheter | Standard Intravenous Non-fenestrated Catheter
Number analyzed (Participants) | 30 | 30
Ratio | 0.72 (0.12) | 0.69 (0.12)

3. Primary Outcome: Image Quality as Assessed by Ratio of Tissue Density of Inferior Vena Cava (IVC) to the Aorta
Description: The ratio of tissue density measured in the inferior vena cava (IVC) to tissue density in the aorta on the CT images will be determined and will provide a measure of biodistribution, which is an important indicator of image quality. Dividing each Hounsfield unit measurement by the aorta density and determining these ratios will be done on a per patient basis to assess biodistribution as a measure of image quality.
Time Frame: at the time of CT scanning
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Becton Dickinson Nexiva Diffusics System Fenestrated Catheter | Standard Intravenous Non-fenestrated Catheter
Number analyzed (Participants) | 31 | 30
Ratio | 0.52 (0.15) | 0.52 (0.18)

4. Primary Outcome: Image Quality as Assessed by Rating Scale
Description: Radiologists blinded to catheter type will review images and rate them on a scale of 1 to 10. 10 indicates a better outcome.
Time Frame: at the time of CT scanning
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Becton Dickinson Nexiva Diffusics System Fenestrated Catheter | Standard Intravenous Non-fenestrated Catheter
Number analyzed (Participants) | 31 | 30
units on a scale | 8.5 (0.97) | 8.6 (0.87)
Statistical Analysis 1: Comparison: Becton Dickinson Nexiva Diffusics System Fenestrated Catheter vs Standard Intravenous Non-fenestrated Catheter; Test type: Superiority; p = 0.4487, two sample t-test

5. Secondary Outcome: Peak Contrast Infusion Pressure
Description: The peak contrast infusion pressure is recorded in the electronic health record (EHR) during every CT examination preformed at the hospitals taking part in this study.
Time Frame: at the time of CT scanning
Population: Peak contrast infusion pressure data was not collected by the technologist for one patient in the "Standard intravenous non-fenestrated catheter" arm.
Measure: Median (Inter-Quartile Range); unit: Pounds per square inch (PSI)
Arm/Group | Becton Dickinson Nexiva Diffusics System Fenestrated Catheter | Standard Intravenous Non-fenestrated Catheter
Number analyzed (Participants) | 31 | 29
Pounds per square inch (PSI) | 80 [71.0 to 89.0] | 93 [81.0 to 114.0]
Statistical Analysis 1: Comparison: Becton Dickinson Nexiva Diffusics System Fenestrated Catheter vs Standard Intravenous Non-fenestrated Catheter; Test type: Superiority; p = 0.0112, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Injection Flow Rate
Description: The injection flow rate is recorded in the electronic health record (EHR) during every CT examination preformed at the hospitals taking part in this study.
Time Frame: at the time of CT scanning
Measure: Mean (Standard Deviation); unit: milliliters per second (mL/sec)
Arm/Group | Becton Dickinson Nexiva Diffusics System Fenestrated Catheter | Standard Intravenous Non-fenestrated Catheter
Number analyzed (Participants) | 31 | 30
milliliters per second (mL/sec) | 2.4 (0.4) | 2.3 (0.3)
Statistical Analysis 1: Comparison: Becton Dickinson Nexiva Diffusics System Fenestrated Catheter vs Standard Intravenous Non-fenestrated Catheter; Test type: Superiority; p = 0.0784, two sample t-test

ADVERSE EVENTS:
Time Frame: 20 minutes after injection of contrast
Description: Every patient was checked for contrast reaction and infiltration of contrast into the skin.
Arm/Group | Becton Dickinson Nexiva Diffusics System Fenestrated Catheter | Standard Intravenous Non-fenestrated Catheter
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 0/31 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes